CLINICAL TRIAL: NCT03467555
Title: Evaluation of Distal Movement of Maxillary Dentition With Zygomatic Miniplates: a Clinical Study Using Cone Beam Computed Tomography
Brief Title: Evaluation of Distal Movement of Maxillary Dentition With Zygomatic Miniplates Using Cone Beam Computed Tomography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sonal tulika
Record Dates: First submitted 2018-03-03; First posted 2018-03-16 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Class II Division 1 Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- distalization group (Experimental): Class II correction using zygomatic miniplates
  Interventions: Device: Class II correction using miniplates in zygomatic region

INTERVENTIONS:
Device: Class II correction using miniplates in zygomatic region

SUMMARY:
The main objective of this study is to quantify the distal movement of maxillary central incisors and molars achieved with miniplate anchorage.

DETAILED DESCRIPTION:
Premolar extraction treatment with multibracketed system and reinforced anchorage has been a common modality for correcting maxillary incisor crowding or Class II malocclusion in nongrowing patients. Treatment of Class II malocclusion without extraction frequently requires distalization of maxillary molars into Class I relation by means of extraoral or intraoral forces. Previously, it had been difficult to move maxillary molars distally after full eruption of maxillary 2nd molars. Extraoral headgear traction restricting the forward growth of maxilla and /or distalizing the maxillary dentition has been the most commonly used and oldest method to correct a Class II buccal segment molar relationship.This distalizes not only 1st molar but also maxillary 1st and 2nd premolars via transeptal fibers. Headgear is seldom an option in adults due to aesthetics and compliance concerns. The disadvantages of extraoral appliances have motivated many investigators to develop the mechanics of intraoral molar distalization.

Various intraoral non compliance appliances like nickel-titanium spring , magnets , distal jet , pendulum appliances have been used to distalize maxillary molars. However, in these appliances, anchorage loss characterized by protrusion of maxillary incisors and an increase in overjet is seen. Also considerable amount of relapse occurred when the distalized molars were used as anchorage for the retraction of anteriors and premolar teeth.

Absolute skeletal anchorage available 24 hours a day is an alternative method for molar distalization. It provides stationary anchorage for various tooth movements without the need for active patient compliance and with no undesirable side effects. Miniscrews, which are generally placed between the roots, limit the amount of distalization possible as they come in contact with surrounding roots during tooth movement. Also, proximity of miniscrews to the roots may lead to failure of screw anchorage .These disadvantages can be overcome by the use of miniplates which are fixed at a distance from the root apices, and therefore do not interfere in tooth movement.

Until now, there have been only a few clinical studies on group distalization of posterior teeth. Thus, little information is available regarding the type of tooth movement that occurs and the limitations of distal movement. An attempt was also not made to study the root resorption and the amount of distal movement or tipping of maxillary 2nd molars since lateral cephalometric radiographs do not provide a clear view of this region.

To the best of our knowledge, no previous study has been conducted on Cone Beam Computed Tomography to evaluate the amount of distal movement of entire maxillary dentition using miniplates placed in zygomatic region and assess the root resorption in all the roots of maxillary molars. The purpose of this study is to evaluate distal movement of maxillary dentition using Cone Beam Computed Tomography to overcome the shortcomings of the previous studies.

MATERIALS AND METHOD Ours is a prospective clinical study to evaluate the distal movement of maxillary dentition achieved in three dimensions with miniplates placed in zygomatic region for the purpose of anchorage. The present study will be conducted in the Department of Orthodontics and Dentofacial Orthopaedics, in conjunction with Department of Oral and Maxillofacial Surgery, P.G.I.D.S., Pt. B.D.Sharma University of Health Sciences, Rohtak. The study will be carried out after the institutional approval obtained from the ethical committee.

SOURCE OF DATA The sample size consists of 20 subjects selected from the patients attending the regular Out Patient Department at the Department of Orthodontics and Dentofacial Orthopaedics for orthodontic treatment.

TARGET SAMPLE SIZE A sample size of 17 for the present study was calculated at 90% power.To compensate for 10% dropouts the final sample size was calculated to be 20.

INTERVENTION AND DESIGN OF STUDY The main intervention in this clinical trial is surgical placement of zygomatic miniplates after initial leveling and alignment of maxillary dental arch. After selection of subjects (patients meeting selection criteria), treatment with 0.022" MBT preadjusted edgewise appliance was started. Maxillary arch will be stabilized with the help of 0.019" × 0.025" stainless steel wire. Pre-treatment diagnostic records and Cone Beam Computed Tomography will be taken before placing miniplates . Maxillary 3rd molars will be extracted, if present . L shaped 2mm titanium miniplates (OrthoMax,Vadodara , India) will be surgically placed under local anaesthesia in aseptic conditions at zygomatic region bilaterally. Hooks will be soldered on archwire used for stabilizing dentition. Ni-Ti closed coil spring/Elastomeric chain will be used to apply a force on both sides (calibrated using Dontrix Gauge ) from miniplates to soldered hooks. Patient will be recalled at 4 weeks interval. Records including Cone Beam Computed Tomography will be taken on achievement of Class I molar relation bilaterally. Lateral cephalograms and CBCT will be taken 2 years post retention.

DATA COLLECTION AND CONE BEAM COMPUTED TOMOGRAPHY ANALYSIS The investigator will record the patients' name, address, contact number and other relevant case history records will be taken. Cephalometric radiographs and Cone Beam Computed Tomography and will be recorded before placement of zygomatic miniplates, on achievement of Class I molar relation bilaterally and 2 years post retention for assessment of distalization. These records will be analyzed. The relevant values will be entered in a predesigned format. Soft tissue profile changes between pretreatment and post treatment will be assessed on lateral cephalogram and the raters- orthodontist, laypersons,patients,parents and general dentists will assess changes in facial appearance on a visual analog scale with profile photographs. Patient perception will be assessed using questionnaire rating by patient regarding various parameters at 1 week, 2 weeks, 1 month and 6 months after the placement of miniplate in zygomatic region. Changes in the upper-airway size will be measured by using lateral cephalometric radiographs taken before and after distalization.

INFORMED CONSENT OF THE PATIENT A valid, informed written consent of the patient or parent/ guardian will be obtained from the patient before registering the patient in this clinical study . Patient will be informed about all the theoretical risks and benefits of the intervention under test .Risks and hazards of radiation during CBCT will also be explained to the patient. The patient will be given 72 hours to discuss the study with his/her family and take the decision regarding participation in the study

ELIGIBILITY:
Inclusion Criteria:

* Non growing patients
* Bilateral Class II molar relationship, defined by at least end-to-end molar relationship.
* No or minor crowding in the mandible.
* Treatment completion without any permanent teeth extracted (excluding third molars).
* Both 1st and 2nd maxillary molars present on the side with a Class II relationship.
* Horizontal to average growth pattern.

Exclusion Criteria:

* Subjects with a history of fixed orthodontic treatment.
* Crossbite
* Vertical growth pattern
* Any systemic disease affecting bone and general growth
* Poor oral hygiene
* Cleft patients
* Patients who fail to follow up or undergo complete treatment

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
distal movement of maxillary molars and central incisors measured in mm at crown and root levels | 24 months
  distal movement of maxillary molars and central incisors before and after intervention measured in mm at crown and root levels on Cone Beam Computed Tomography
root resorption of maxillary teeth | 24 months
  root resorption of maxillary incisors, canines, premolars and molars evaluated by measuring the root lengths along the long axis of the roots from cemento- enamel junction to the root tips in mm on Cone Beam Computed Tomography before and after intervention
patient experiences with zygomatic miniplates | 20 months
  questionaires given to patients for evaluating patient attitude and pain perception (using Visual Analog Scale) at different time intervals.
soft tissue profile changes | 30 months
  soft tissue profile changes after intervention evaluated on lateral cephalogram and the raters- orthodontist, laypersons,patients,parents and general dentists will assess changes in facial appearance on a visual analog scale with profile photographs

SECONDARY OUTCOMES:
mandibular plane angle | 24 months
  changes in mandibular plane angle after intervention
the movement of maxillary central incisors and molars in vertical plane | 24 months
  the movement of maxillary central incisors and molars in vertical plane assessed by measuring the perpendicular distance between the incisal edge/ mesio-buccal cusp to the palatal plane on Cone Beam Computed Tomography
transverse changes | 24 months
  intercanine and intermolar width will be assessed on CBCT before and after distalization
Airway changes | 24 months
  changes in the upper-airway size will be measured by using lateral cephalometric radiographs before and after distalization

CONTACTS AND LOCATIONS:
Overall Officials: Sonal Chowdhary, Principal Investigator — POST GRADUATE INSTITUTE OF DENTAL SCIENCES
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol